CLINICAL TRIAL: NCT00002907
Title: PHASE II CLINICAL EVALUATION OF BRYOSTATIN 1 IN PATIENTS WITH RELAPSED MULTIPLE MYELOMA
Brief Title: Bryostatin 1 in Treating Patients With Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065272; P30CA022453 (NIH); WSU-C-1257; WSU-D-1257; NCI-T95-0062D
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — bryostatin 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bryostatin 1

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of bryostatin 1 in treating patients with relapsed multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of bryostatin 1 administered as a 72-hour continuous infusion in patients with relapsed multiple myeloma. II. Determine the qualitative and quantitative toxic effects of bryostatin 1 in these patients. III. Determine the duration of response and survival following bryostatin 1 in these patients.

OUTLINE: All patients receive bryostatin 1 by 72-hour continuous infusion every 2 weeks until disease progression or 2 courses beyond complete remission. Response is assessed after every 4 courses. Patients are followed for survival.

PROJECTED ACCRUAL: A total of 15-25 evaluable patients will be entered into this study over 1.25 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Multiple myeloma of any stage that has failed 1 or 2 prior regimens (chemotherapy, biologic therapy, or both, or bone marrow transplantation) Evidence of disease progression required Ineligible for known treatment of higher potential efficacy One of the following protein criteria required: Quantifiable M-components of IgG, IgA, IgD, or IgE Urinary kappa or lambda light chain (Bence-Jones protein) excretion Re-treatment on this protocol allowed if disease relapsed after a complete remission

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 50,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL Transaminases less than 2.5 times normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No history of impaired cardiac status, e.g.: Severe coronary artery disease Cardiomyopathy Congestive heart failure Arrhythmia Other: No known AIDS or HIV infection No second malignancy within 5 years except: Adequately treated nonmelanomatous skin cancer Carcinoma in situ of the cervix No pregnant or nursing women Effective contraception required of fertile patients during and for 2 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics At least 4 weeks since chemotherapy (8 weeks since mitomycin or nitrosoureas) and recovered Endocrine therapy: No concurrent steroids Radiotherapy: At least 4 weeks since radiotherapy and recovered Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-01; Primary Completion 1999-01 (Actual); Study Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayad M. Al-Katib, MD, FACP, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States